CLINICAL TRIAL: NCT02087982
Title: Development of General Practitioners Screening Tool of Frail Older Old Community-dwellers: a Cohort Population-based Study
Brief Title: Development of General Practitioners Screening Tool of Frail Older Old Community
Acronym: ReperAge
Status: Completed | Type: Observational
Sponsor: Gerontopôle des Pays de la Loire (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: Reperage - 23
Record Dates: First submitted 2013-10-28; First posted 2014-03-14 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Aged (80 or More); Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Seniors: The study will be based on a 6-months assessment period, with two consecutive monitoring visits on enrollment.
  Patient follow-up after 3 months will be conducted by telephone and monitoring after 6 months will be carried out as part of a routine consultation.
  Each subject will have a BGA (Brief Geriatric assesment).

SUMMARY:
The comprehensive geriatric assessment (CGA) is a multidimensional, interdisciplinary diagnostic process to determine the medical, psychological, and functional capabilities of an elderly person, in order to develop a coordinated and integrated plan for treatment. It represents the first stage of the most appropriate care for elderly people who are frail or who cannot perform at least three daily tasks unaided.

It has been shown that the integration of CGA in the decision-making and care management at hospital improves inpatient's health and functional status, and reduces mortality rate and healthcare expenditures. The effects of CGA in daily practice of general practitioners remain unknown.

Implementation of a systematic CGA for every older old community-dwellers performed by a general practitioner remains yet difficult because of number of issues. First, although the number of older old community-dwellers keeps increasing, the number of health care professional with geriatric skills does not. Second, CGA is a complex and time-consuming process. Third, CGA requires a multidisciplinary geriatric team that cannot support alone the care of all frail older old community-dwellers due to their limited number. An implication of non-geriatricians in CGA is therefore required.

Recently, it was confirmed that CGA cannot be applied to all older adults, and that the best compromise could be the use of a two-step approach. The first step is the identification by non-geriatricians of elderly inpatients at high risk of adverse outcomes using a screening tool, and the second step is a CGA by geriatricians with a diagnosis purpose.

None of existing tools used for screening is adapted to the population of elderly people who visit general practitioners.Thus, healthcare professionals working in ED need a simple, standardized and brief geriatric assessment (BGA) to identify as soon as possible frail older old community-dwellers requiring specialized geriatric care.

The investigators hypothesized that a BGA older old community-dwellers carried out by a general practitioner could predict the adverse health events (i.e. hospitalization, institutionalisation, medical consultations and death) occurring during a 6-months follow-up period before the evaluation.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are those who meet the following inclusion criteria:

* the patient is aged 80 or more,
* the patient comes to a normal medical consultation without any acute health problem,
* the patient lives at home,
* the patient is able to respond to questions he is asked,
* the patient has given his agreement to answer questions during the initial consultation, to answer further questions by telephone after 3 months and to return in 6 months for a further consultation,
* the life expectancy of the patient as estimated by the primary care practitioner is greater than 6 months.
* the patient has french nationality and is a member of a national Social Security scheme.

Exclusion Criteria:

Patients are ineligible if :

* one inclusion criteria is not met,
* if a close relation of the patient does not agree the patient to be part of the study.

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: adults aged 80 and over
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of non planned hospitalization by subjects | Hospitalization between inclusion and follow up to 6 months
  The BGA test will include the following criteria:
  * age,
  * sex,
  * the ability to give the current month and year,
  * the occurrence of falls during the last 6 months,
  * the presence of more than 4 classes of prescribed drugs,
  * the presence of professional or other assistance help at home.
  All following adverse health events occurring during a 6-months period of follow-up :
  * Hospitalization,
  * Institutionalisation,
  * Medical consultations,
  * Death.

SECONDARY OUTCOMES:
Number of subjects' institutionnalized | Institutionnalization between inclusion and follow up at 3 or 6 months
Number of dead subjects | Death between inclusion and follow up at 3 or 6 months

OTHER OUTCOMES:
Number of non planned consultations by subjects | Number of non planned consultations between inclusion and follow up at 3 or 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Berrut, PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nord Pas de Calais, Leers, France